CLINICAL TRIAL: NCT01996267
Title: Optimizing Neoadjuvant Systemic Treatment for HER2 Positive Breast Cancer - the TRAIN-2 Study
Brief Title: Neoadjuvant Chemotherapy in HER2 Positive Breast Cancer, TRAIN-2
Acronym: TRAIN-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Roche Pharma AG (Industry); Borstkanker Onderzoek Groep (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13TRT
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; HER2 Positive
Keywords: neoadjuvant; breast cancer; HER2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; Carboplatin; pertuzumab; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FEC-T +Pertuzumab (Active Comparator): Fluorouracil; 500 mg/m2; day 1 Epirubicine; 90 mg/m2; day 1 Cyclophosphamide; 500 mg/m2; day 1 Trastuzumab; 6 mg/kg (loading dose 8 mg/kg) Pertuzumab; 420 mg (loading dose 840 mg); day 1 Cycle is repeated every 21 days
  Interventions: Drug: FEC-T+Pertuzumab
- PTC+Pertuzumab (Active Comparator): Paclitaxel; 80 mg/m2; day 1,8 Trastuzumab; 6 mg/kg (loading dose 8 mg/kg); day 1 Carboplatin; AUC=6; day 1 Pertuzumab; 420 mg (loading dose 840 mg); day 1 Cycle repeated every 21 days
  Interventions: Drug: PTC+Pertuzumab

INTERVENTIONS:
Drug: PTC+Pertuzumab — Cycle repeated every 21 days
  Other Names: Paclitaxel; 80 mg/m2; day 1,8; Trastuzumab; 6 mg/kg (loading dose 8 mg/kg); day 1; Carboplatin; AUC=6; day 1; Pertuzumab; 420 mg (loading dose 840 mg); day 1
  Arms: PTC+Pertuzumab
Drug: FEC-T+Pertuzumab — Cycle is repeated every 21 days
  Other Names: Fluorouracil; 500 mg/m2; day 1; Epirubicine; 90 mg/m2; day 1; Cyclophosphamide 500 mg/m2; day 1; Trastuzumab; 6 mg/kg (loading dose 8 mg/kg); Pertuzumab; 420 mg (loading dose 840 mg); day 1
  Arms: FEC-T +Pertuzumab

SUMMARY:
This study compares two schedules of upfront chemotherapy in HER positive breast cancer.

DETAILED DESCRIPTION:
Upfront trastuzumab treatment is beneficial to patients with HER2 positive breast cancer. The potential synergistic cardiotoxicity of trastuzumab and anthracyclines has led to the development of non-anthracycline containing regimens, which have shown high pathologic complete response rates. Anthracyclines remain very active in HER2 positive breast cancer, however, and increasing evidence now supports safe combination of trastuzumab and epirubicin. Therefore, the addition of epirubicin to a non-anthracycline containing regimen may further improve outcome for patients with HER2 positive breast cancer.

Several reports confirmed benefit of dual HER2 blockade by adding pertuzumab to a trastuzumab containing neoadjuvant regimen. The results of the combined treatment in the Neosphere study, however, are similar to what we found in a phase II trial using a weekly paclitaxel, trastuzumab, carboplatin combination with pCR rates of approximately 44%. Adding pertuzumab to this regimen is likely to also increase the high pCR rate and to add substantial benefit to patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed infiltrating breast cancer
* Stage II or stage III disease. Nodal status must be examined by ultrasound, fine needle aspiration, sentinel node biopsy, or FDG-PET scan.
* Overexpression and/or amplification of HER2 in an invasive component of the core biopsy, according to one of the following definitions:

  •>30% of invasive tumor cells showing strong complete circumferential membrane staining (score 3+)

  •HER2 gene amplification defined as >6 HER2 gene copies per nucleus by in situ hybridization.
* Age ≥18
* Eastern Cooperative Oncology Group performance status ≤1
* Adequate bone marrow function (ANC >1.5 x 109/l, platelets >100 x 109/l)
* Adequate hepatic function (ALAT, ASAT and bilirubin <2.5 times upper limit of normal)
* Adequate renal function (creatinine clearance >50 ml/min)
* LVEF ≥50% measured by echocardiography or MUGA
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Absence of any medical condition that would place the patient at unusual risk.
* Signed written informed consent

Exclusion Criteria:

* previous radiation therapy or chemotherapy
* other malignancy except carcinoma in situ, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiation therapy.
* current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection
* evidence of distant metastases. Evaluation of the presence of distant metastases may include chest X-ray, liver ultrasound, isotope bone-scan, CT-scan of chest and abdomen and/or FDG-PET scan, according to local procedures.
* evidence of bilateral infiltrating breast cancer. Evaluation of the presence of bilateral infiltrating breast cancer may include mammography, breast ultrasound and/or MRI breast.
* concurrent anti-cancer treatment or another investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2013-12; Primary Completion 2018-12 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pathological complete response | at week 30
  To compare the efficacy of six cycles neoadjuvant PTC plus pertuzumab preceded by either three cycles of FEC-T plus pertuzumab or three cycles of PTC plus pertuzumab in HER2 positive breast cancer

SECONDARY OUTCOMES:
Number of patients with grade >2 adverse events as a measure of safety and tolerability | up to week 35
  to describe the safety of the various regimens toxicity is compared between the two arms
identify prognostic and predictive biomarkers for pCR | within one year after end of treatment
  To identify prognostic and predictive biomarkers for pCR after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gabe S Sonke, MD, Principal Investigator — Antoni van Leeuwenhoek, Amsterdam
Locations (33):
- Netherlands (33):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - MCA, Alkmaar
  - ZGT, Almelo
  - Antoni van Leeuwenhoek, Amsterdam
  - AZVU, Amsterdam
  - OLVG, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Deventer ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - St Anna Geldrop, Geldrop
  - Orbis Medisch Centrum, Geleen
  - Groene Hart, Gouda
  - Kennemer Gasthuis, Haarlem
  - Atrium Medisch Centrum Parkstad, Heerlen
  - Spaarne ziekenhuis, Hoofddorp
  - Westfries Gasthuis, Hoorn
  - MCL, Leeuwarden
  - LUMC, Leiden
  - Diaconessenhuis Meppel, Meppel
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Waterlandziekenhuis, Purmerend
  - Vlietland Ziekenhuis, Schiedam
  - Haga, The Hague
  - Bronovo Ziekenhuis, The Hague
  - St. Elisabeth, Tilburg
  - Diaconessenhuis Utrecht, Utrecht
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo
  - Zaans Medisch Centrum, Zaandam
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] van der Voort A, van Ramshorst MS, van Werkhoven ED, Mandjes IA, Kemper I, Vulink AJ, Oving IM, Honkoop AH, Tick LW, van de Wouw AJ, Mandigers CM, van Warmerdam LJ, Wesseling J, Vrancken Peeters MT, Linn SC, Sonke GS. Three-Year Follow-up of Neoadjuvant Chemotherapy With or Without Anthracyclines in the Presence of Dual ERBB2 Blockade in Patients With ERBB2-Positive Breast Cancer: A Secondary Analysis of the TRAIN-2 Randomized, Phase 3 Trial. JAMA Oncol. 2021 Jul 1;7(7):978-984. doi: 10.1001/jamaoncol.2021.1371. PMID 34014249
- [Derived] van Ramshorst MS, van der Voort A, van Werkhoven ED, Mandjes IA, Kemper I, Dezentje VO, Oving IM, Honkoop AH, Tick LW, van de Wouw AJ, Mandigers CM, van Warmerdam LJ, Wesseling J, Vrancken Peeters MT, Linn SC, Sonke GS; Dutch Breast Cancer Research Group (BOOG). Neoadjuvant chemotherapy with or without anthracyclines in the presence of dual HER2 blockade for HER2-positive breast cancer (TRAIN-2): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2018 Dec;19(12):1630-1640. doi: 10.1016/S1470-2045(18)30570-9. Epub 2018 Nov 6. PMID 30413379